CLINICAL TRIAL: NCT03456557
Title: The Use of Perfusion CT Derived Parameters as Early Acute Pancreatitis Severity Biomarker Compared to Clinico Biological Score
Acronym: K-PA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K-PA Study
Record Dates: First submitted 2018-02-22; First posted 2018-03-07 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Cytidine Triphosphate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computed tomography. (Experimental)
  Interventions: Radiation: Perfusion computed tomography.

INTERVENTIONS:
Radiation: Perfusion computed tomography. — Using specific post treatment imaging software ( Olea® ) we will calculatell permeability parameters : the pancreatic blood flow and the k-trans, capillary membrane permeability factor.

SUMMARY:
The investigators to establish whether early microvascular permeability parameter evaluated by perfusion-CT could be good biomarkers for severity in acute pancreatitis.

Therefore the investigators want to compare 48 hours-clinico-biological systemic inflammatory response syndrome score to initial microvascular permeability parameters ( ktrans - capillary membrane permeability factor- and pancreatic blood flow ) calculated by OLEA software using inclusion perfusion CT.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acute pancreatitis (based on the Atlanta definition).

Exclusion Criteria:

* Patient under 18 yearras old
* Contraindication of injection of iodinated contrast medium
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-12-09 (Actual); Study Completion 2018-12-09 (Actual)

PRIMARY OUTCOMES:
Relation between CT perfusion calculated k-trans and clinicobiological SIRS score in early phase of acute pancreatitis. | admission day

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Poitiers, Poitiers, France